CLINICAL TRIAL: NCT05402007
Title: Clinical and Functional Effects of Supervised and Unsupervised Cardiopulmonary Rehabilitation in POST-COVID-19 Syndrome: Clinical and Randomized Trial
Brief Title: Effects of Cardiopulmonary Rehabilitation in Participants With Post-COVID 19 Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Ana Carolina Sebastião da Silva, Master's Degree, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTC20457
Record Dates: First submitted 2022-04-06; First posted 2022-06-02 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Post- COVID-19 Syndrome; Exercises; Pulmonary Rehabilitation; COVID-19; Randomized Clinical Trial
Keywords: COVID-19; Post- COVID-19 syndrome; Pulmonary Rehabilitation; Exercises
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity; COVID-19

STUDY DESIGN:
Intervention Model Description: Three pre-post assessment groups (control/face-to-face intervention/self-performed home intervention)
Who Masked: Investigator
Masking Description: The study will be a clinical trial previously randomized by electronic randomization system (www.random.org) and the allocation of volunteers in the study arms will be done without the participation of the researchers. The study will be double-blind since neither the volunteers nor the professional who will perform the Cardiopulmonary Rehabilitation protocol is aware of the objectives and clinical valences that will be measured by the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group will not receive intervention during the study.
- Face-to-face intervention (Active Comparator): The face-to-face intervention group will perform pulmonary rehabilitation at the professional-oriented Rehabilitation Center.
  Interventions: Other: Pulmonary rehabilitation exercises at the Rehabilitation Center
- Home intervention (Active Comparator): The home intervention group will carry out home intervention through a self-explanatory exercise booklet.
  Interventions: Other: Home Intervention

INTERVENTIONS:
Other: Pulmonary rehabilitation exercises at the Rehabilitation Center — Face-to-face intervention (12 weeks): Using the participants' assessment and personal characteristics, the therapist will prescribe pulmonary rehabilitation exercises that will be performed at the pulmonary rehabilitation center.
  Arms: Face-to-face intervention
Other: Home Intervention — Home Intervention (12 weeks): Using the participants' assessment and personal characteristics, the therapist will provide a portfolio of self-explanatory exercises, and guide participants on safety precautions.
  Arms: Home intervention

SUMMARY:
COVID-19 is an emerging pandemic disease caused by severe acute respiratory syndrome (SARS-CoV-2). Although the majority of patients infected with SARS-CoV-2 are asymptomatic or have mild symptoms, some patients develop severe symptoms that can protractedly impair their quality of life and functional capacity. SARS-CoV-2 is closely related to severe acute respiratory syndrome (SARS) with direct and indirect effects on several systems, especially the musculoskeletal system, in addition to the respiratory system. Some of these symptoms persist for a long period, called Post-Covid-19 Syndrome, directly interfering with the functional capacity and quality of life of these participants. Cardiopulmonary Rehabilitation exercises are focused on restoring functional capacity in patients affected by cardiopulmonary diseases. The primary objective of this study is to evaluate the clinical and functional effects of a quarterly Cardiopulmonary Rehabilitation exercise program for participants with post-COVID-19 syndrome.

The secondary objectives will be: To compare the effects of a supervised program of 12 weeks of supervised exercises and a program of self-performed home exercises, guided by an exercise booklet, of the same duration on muscle strength and peripheral resistance; Compare the effects of a 12-week supervised exercise program and a self-performed home exercise program, guided by an exercise booklet, of the same duration on levels of fatigue and dyspnea in patients with post-COVID-19 syndrome; Compare the effects of a 12-week supervised exercise program and a self-performed home exercise program, guided by an exercise booklet, of the same duration on health-related quality of life and post-COVID-19 functional status.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blind treatment trial with a 1:1 allocation ratio.

Participants: Patients will be recruited at the Central Hospital of the Military Police and in the specialized multidisciplinary follow-up outpatient clinic after COVID-19. The participants will be adults (≥18 years and ≤ 65 years), with a previous diagnosis COVID-19, who required hospitalization and need for invasive mechanical ventilation for at least 7 days and who were discharged from the hospital between August and Dec 2021.

Intervention and comparison:

This study will be divided into three groups: control group, face-to-face intervention group and home intervention group. Both groups will be evaluated before and after the study period, however the control group will only receive the treatment offered to the other groups after the end of the study. Physical functions and functional capacity will be evaluated.

After ensuring that patients meet the inclusion criteria, they will be divided into groups that will receive supervised care in a supervised Pulmonary Rehabilitation Center, with protocoled exercises, the other group will receive a booklet of self-explanatory exercises for performing the exercises in home, and the control group that will not receive intervention in this period.

The intervention groups should perform the exercises in the period of 12 weeks, 2 times a week, totaling 24 intervention sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with COVID-19, who required hospitalization and required invasive mechanical ventilation for at least 7 days and who were discharged between August and December 2021 to minimize regression to mean;
* Both sexes;
* Over 18 years old and under 65 years old.

Exclusion Criteria:

* Need for supplemental home oxygen;
* Motor or neurological or cognitive alteration that contraindicates the participation in the cardiopulmonary rehabilitation program.
* Persistence of clinical signs of deep vein thrombosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Peripheral muscle function I | 12 weeks
  Will be assessed using the Palm Grip Dynamometry
Peripheral muscle function II | 12 weeks
  Will be assessed using the Quadriceps Peak Load Test
Peripheral muscle function III | 12 weeks
  Will be assessed using the Quadriceps Muscle Endurance Test.
Daily living activity | 12 weeks
  It will be evaluated by the modified Medical Resource Council (mMRC) dyspnea scale

SECONDARY OUTCOMES:
Quality of life improvement | 12 weeks
  The assessment of quality of life will be carried out using a generic instrument of 36 items, validated in Brazil and called the SF-36 (Short Form Health Survey).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina Sebastião da Silva, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro de Fisiatria e Reabilitação da Polícia Militar- RJ, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No